CLINICAL TRIAL: NCT04537208
Title: Immunogenicity and Safety of SARS-CoV-2 Recombinant Protein Vaccine Formulations (With or Without Adjuvant) in Healthy Adults 18 Years of Age and Older
Brief Title: Study of Recombinant Protein Vaccine Formulations Against COVID-19 in Healthy Adults 18 Years of Age and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAT00001; U1111-1250-4757 (Other: UTN)
Record Dates: First submitted 2020-09-02; First posted 2020-09-03 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 (Healthy Volunteers)
MeSH Terms: conditions — COVID-19 | interventions — Adjuvants, Pharmaceutic; Saline Solution

STUDY DESIGN:
Intervention Model Description: This was a parallel group prevention study. Participants from 2 age groups (adults 18 through 49 years of age and adults 50 years of age and older) received either 1 injection (Cohort 1) or 2 injections (Cohort 2) of study vaccine or placebo control.
  As a precautionary step, a sentinel safety cohort of 6 participants (younger adults only) within each dosing group from Cohort 1 was enrolled. An early safety data review was performed, including evaluation of safety data and laboratory measures to Day 9. Upon acceptable safety demonstrated from unblinded data review by limited members of the Sponsor Study Team, the remaining participants were enrolled simultaneously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, outcome assessors, Investigators, laboratory personnel, and the majority of Sponsor study staff will be blinded to vaccine group assignment; injection schedule will be unblinded and those preparing/administering the study interventions will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort 1: Group 1: SARS-CoV-2 vaccine LD + AF03 (Experimental): Participants received a single intramuscular (IM) injection of SARS-CoV2 vaccine low-dose (LD) formulation along with adjuvant AF03 on Day 1.
  Interventions: Biological: CoV2 preS dTM-AF03 (low-dose)
- Cohort 1: Group 2: SARS-CoV-2 vaccine LD + AS03 (Experimental): Participants received a single IM injection of SARS-CoV2 vaccine LD formulation along with adjuvant AS03 on Day 1.
  Interventions: Biological: CoV2 preS dTM-AS03 (low-dose)
- Cohort 1: Group 3: SARS-CoV-2 vaccine HD + AF03 (Experimental): Participants received a single IM injection of SARS-CoV2 vaccine high-dose (HD) formulation along with adjuvant AF03 on Day 1.
  Interventions: Biological: CoV2 preS dTM-AF03 (high-dose)
- Cohort 1: Group 4: SARS-CoV-2 vaccine HD + AS03 (Experimental): Participants received a single IM injection of SARS-CoV2 vaccine HD formulation along with adjuvant AS03 on Day 1.
  Interventions: Biological: CoV2 preS dTM-AS03 (high-dose)
- Cohort 1: Group 5: Placebo (Placebo Comparator): Participants received an IM injection of placebo matching to SARS-CoV2 vaccine on Day 1.
  Interventions: Biological: Placebo (0.9% normal saline)
- Cohort 2: Group 6: SARS-CoV-2 vaccine LD + AF03 (Experimental): Participants received IM injection of SARS-CoV2 vaccine LD formulation along with adjuvant AF03 on Day 1 and Day 22, respectively.
  Interventions: Biological: CoV2 preS dTM-AF03 (low-dose)
- Cohort 2: Group 7: SARS-CoV-2 vaccine LD + AS03 (Experimental): Participants received IM injection of SARS-CoV2 vaccine LD formulation along with adjuvant AS03 on Day 1 and Day 22, respectively.
  Interventions: Biological: CoV2 preS dTM-AS03 (low-dose)
- Cohort 2: Group 8: SARS-CoV-2 vaccine HD + AF03 (Experimental): Participants received IM injection of SARS-CoV2 vaccine HD formulation along with adjuvant AF03 on Day 1 and Day 22, respectively.
  Interventions: Biological: CoV2 preS dTM-AF03 (high-dose)
- Cohort 2: Group 9: SARS-CoV-2 vaccine HD + AS03 (Experimental): Participants received IM injection of SARS-CoV2 vaccine HD formulation along with adjuvant AS03 on Day 1 and Day 22, respectively.
  Interventions: Biological: CoV2 preS dTM-AS03 (high-dose)
- Cohort 2: Group 10: SARS-CoV-2 vaccine HD (Experimental): Participants received a single IM injection of SARS-CoV2 vaccine HD formulation without adjuvant on Day 1 and Day 22, respectively.
  Interventions: Biological: CoV2 preS dTM (high-dose) without adjuvant
- Cohort 2: Group 11: Placebo (Placebo Comparator): Participants received an IM injection of placebo matching to SARS-CoV2 on Day 1 and Day 22, respectively.
  Interventions: Biological: Placebo (0.9% normal saline)

INTERVENTIONS:
Biological: CoV2 preS dTM-AF03 (low-dose) — Pharmaceutical form: liquid; route of administration: intramuscular injection
  Arms: Cohort 1: Group 1: SARS-CoV-2 vaccine LD + AF03; Cohort 2: Group 6: SARS-CoV-2 vaccine LD + AF03
Biological: CoV2 preS dTM-AF03 (high-dose) — Pharmaceutical form: liquid; route of administration: intramuscular injection
  Arms: Cohort 1: Group 3: SARS-CoV-2 vaccine HD + AF03; Cohort 2: Group 8: SARS-CoV-2 vaccine HD + AF03
Biological: CoV2 preS dTM-AS03 (low-dose) — Pharmaceutical form: liquid; route of administration: intramuscular injection
  Arms: Cohort 1: Group 2: SARS-CoV-2 vaccine LD + AS03; Cohort 2: Group 7: SARS-CoV-2 vaccine LD + AS03
Biological: CoV2 preS dTM-AS03 (high-dose) — Pharmaceutical form: liquid; route of administration: intramuscular injection
  Arms: Cohort 1: Group 4: SARS-CoV-2 vaccine HD + AS03; Cohort 2: Group 9: SARS-CoV-2 vaccine HD + AS03
Biological: CoV2 preS dTM (high-dose) without adjuvant — Pharmaceutical form: liquid; route of administration: intramuscular injection
  Arms: Cohort 2: Group 10: SARS-CoV-2 vaccine HD
Biological: Placebo (0.9% normal saline) — Pharmaceutical form: liquid; route of administration: intramuscular injection
  Arms: Cohort 1: Group 5: Placebo; Cohort 2: Group 11: Placebo

SUMMARY:
The primary objectives of the study were:

* To describe the neutralizing antibody profile at Day 1, Day 22, and Day 36 of each study intervention group.
* To describe the safety profile of all participants in each age group and each study intervention group up to 12 months post-last injection.

The secondary objectives of the study are:

* To describe binding antibody profile at Day 1, Day 22, Day 36, Day 181 (Cohort 1) or Day 202 (Cohort 2), and Day 366 (Cohort 1) or Day 387 (Cohort 2) of each study intervention group.
* To describe the neutralizing antibody profile at Day 181 (Cohort 1) or Day 202 (Cohort 2) and at Day 366 (Cohort 1) and Day 387 (Cohort 2) of each study intervention group.
* To describe the occurrence of virologically-confirmed coronavirus disease (COVID-19)-like illness and serologically-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* To evaluate the correlation / association between antibody responses to SARS-CoV-2 Recombinant Protein and the risk of virologically-confirmed COVID-19-like illness and/or serologically-confirmed SARS-CoV-2 infection.

DETAILED DESCRIPTION:
The duration of each participant's participation in the study was approximately 365 days (Cohort 1) and 386 days (Cohort 2) post last injection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or older on the day of inclusion.
* Informed consent form had been signed and dated.
* Able to attend all scheduled visits and complied with all study procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not used an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 12 weeks after the last vaccination. To be considered of non-childbearing potential, a female was post-menopausal for at least 1 year or surgically sterile.
* Receipt of any vaccine in the 30 days preceding the first study vaccination or planned receipt of any vaccine in the 30 days following the last study vaccination except for influenza vaccination, which might be received at least 2 weeks before and a minimum of 2 weeks after study vaccines.
* Prior administration of a coronavirus vaccine SARS-CoV-2, SARS-CoV, Middle East Respiratory Syndrome).
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of SARS-CoV-2 infection, confirmed either clinically, serologically, or microbiologically
* Chronic illness or condition considered to potentially increase the risk for severe COVID illness or that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Receipt of any therapy known to had in-vitro antiviral activity against SARS-CoV-2 within 72 hours prior to the first blood drew.
* Health care workers provided direct participant care for COVID-19 participants.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (11):
- United States (11):
  - Investigational Site Number 8400004, Birmingham, Alabama
  - Investigational Site Number 8400012, Rolling Hills Estates, California
  - Investigational Site Number 8400011, Hollywood, Florida
  - Investigational Site Number 8400019, Melbourne, Florida
  - Investigational Site Number 8400016, Boston, Massachusetts
  - Investigational Site Number 8400002, Omaha, Nebraska
  - Investigational Site Number 8400001, Rochester, New York
  - Investigational Site Number 8400007, Rochester, New York
  - Investigational Site Number 8400008, Cleveland, Ohio
  - Investigational Site Number 8400003, Philadelphia, Pennsylvania
  - Investigational Site Number 8400014, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] De Rosa SC, Cohen KW, Bonaparte M, Fu B, Garg S, Gerard C, Goepfert PA, Huang Y, Larocque D, McElrath MJ, Morris D, Van der Most R, de Bruyn G, Pagnon A. Whole-blood cytokine secretion assay as a high-throughput alternative for assessing the cell-mediated immunity profile after two doses of an adjuvanted SARS-CoV-2 recombinant protein vaccine candidate. Clin Transl Immunology. 2022 Jan 11;11(1):e1360. doi: 10.1002/cti2.1360. eCollection 2022. PMID 35035955
- [Derived] Goepfert PA, Fu B, Chabanon AL, Bonaparte MI, Davis MG, Essink BJ, Frank I, Haney O, Janosczyk H, Keefer MC, Koutsoukos M, Kimmel MA, Masotti R, Savarino SJ, Schuerman L, Schwartz H, Sher LD, Smith J, Tavares-Da-Silva F, Gurunathan S, DiazGranados CA, de Bruyn G. Safety and immunogenicity of SARS-CoV-2 recombinant protein vaccine formulations in healthy adults: interim results of a randomised, placebo-controlled, phase 1-2, dose-ranging study. Lancet Infect Dis. 2021 Sep;21(9):1257-1270. doi: 10.1016/S1473-3099(21)00147-X. Epub 2021 Apr 19. PMID 33887209
- See also: VAT00001 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25373&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 active sites in the United States between 03 September 2020 to 19 November 2021.
Pre-assignment Details: A total of 441 participants were enrolled, of which 439 were vaccinated in the study.
Groups:
- Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03: Participants received a single intramuscular (IM) injection of severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccine low-dose (LD) formulation along with adjuvant AF03 on Day 1.
- Cohort 1: Group 5: Placebo: Participants received a single IM injection of placebo matching to SARS-CoV2 vaccine on Day 1.
- Cohort 2: Group 10: SARS-CoV-2 Vaccine HD: Participants received IM injection of SARS-CoV2 vaccine HD formulation without adjuvant on Day 1 and Day 22, respectively.
- Cohort 2: Group 11: Placebo: Participants received IM injection of placebo matching to SARS-CoV2 vaccine on Day 1 and Day 22, respectively.
Period: Overall Study
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Started | 34 | 34 | 34 | 34 | 34 | 28 | 84 | 27 | 85 | 18 | 29
Vaccinated on Day 1 | 34 | 34 | 34 | 34 | 34 | 28 | 82 | 27 | 85 | 18 | 29
Vaccinated on Day 22 (Only Cohort 2 participants received second dose of vaccine at Day 22.) | 0 | 0 | 0 | 0 | 0 | 26 | 80 | 26 | 85 | 17 | 29
Safety Analysis Set (SafAS) (Participants who had received at least one injection of study intervention and were analyzed according to the study intervention they actually received.) | 36 (2 participants randomized to 'Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03' received only one injection in Cohort 2 and thus included in arm 'Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03' for safety analysis.) | 36 (2 participants randomized to 'Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03' received only one injection in Cohort 2 and thus included in arm 'Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03' for safety analysis.) | 35 (1 participant randomized to 'Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03' received only one injection in Cohort 2 and thus included in arm 'Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03' for safety analysis.) | 34 | 34 | 26 (2 participants randomized to 'Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03' received only one injection in Cohort 2 and thus included in arm 'Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03' for safety analysis.) | 80 (2 participants randomized to 'Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03' received only one injection in Cohort 2 and thus included in arm 'Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03' for safety analysis.) | 26 (1 participant randomized to 'Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03' received only one injection in Cohort 2 and thus included in arm 'Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03' for safety analysis.) | 85 | 18 | 29
Completed | 26 | 31 | 28 | 27 | 26 | 23 | 71 | 24 | 69 | 14 | 21
Not Completed | 8 | 3 | 6 | 7 | 8 | 5 | 13 | 3 | 16 | 4 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 2 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 3 | 5 | 1 | 6 | 1 | 7 | 2 | 4
Not completed — Lost to Follow-up | 4 | 1 | 3 | 4 | 3 | 2 | 3 | 2 | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03: Participants received a single IM injection of SARS-CoV2 vaccine LD formulation along with adjuvant AF03 on Day 1.
- Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03: Participants received a single IM injection of SARS-CoV2 vaccine HD formulation along with adjuvant AF03 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo | Total
Number analyzed (Participants) | 34 | 34 | 34 | 34 | 34 | 28 | 84 | 27 | 85 | 18 | 29 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (14.2) | 41.9 (12.8) | 39.8 (15.5) | 39.0 (17.2) | 39.6 (15.7) | 43.7 (14.1) | 42.9 (14.9) | 42.2 (15.5) | 44.7 (15.5) | 34.8 (10.2) | 43.2 (16.2) | 42.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 17 | 21 | 18 | 14 | 36 | 18 | 44 | 10 | 14 | 229
  Male | 12 | 19 | 17 | 13 | 16 | 14 | 48 | 9 | 41 | 8 | 15 | 212
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Asian | 2 | 3 | 1 | 5 | 1 | 3 | 7 | 0 | 4 | 1 | 1 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 1 | 0 | 1 | 0 | 1 | 4 | 1 | 3 | 1 | 2 | 15
  White | 29 | 28 | 30 | 25 | 30 | 24 | 72 | 25 | 78 | 16 | 26 | 383
  More than one race | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5
  Unknown or Not Reported | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine Formulations at Day 1
Description: GMTs of SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. Titers were expressed in terms of 1/dilution.
Time Frame: Day 1 (pre-vaccination)
Population: Analysis was performed on Per-protocol analysis set for immunogenicity (PPAS-IAS) population which included all participants who received at least one injection of study intervention and had evaluable immunogenicity data, with no major protocol violations. Here, "overall number of participants analyzed" signifies participants with available data for this outcome measure (OM).
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 21 | 20 | 24 | 25 | 17 | 67 | 22 | 68 | 13 | 22
titers | 5.00 [NA to NA] — 95% confidence interval (CI) was not computable as the standard deviation (SD) of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

2. Primary Outcome: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine Formulations at Day 22
Description: as for outcome 1
Time Frame: Day 22 (post-vaccination)
Population: Analysis was performed on PPAS-IAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 18 | 68 | 22 | 69 | 13 | 22
titers | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.27 [4.72 to 5.89] | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.29 [4.89 to 5.73] | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.59 [4.93 to 6.34] | 5.35 [4.62 to 6.19] | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

3. Primary Outcome: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine Formulations at Day 36
Description: as for outcome 1
Time Frame: Day 36 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 17 | 60 | 20 | 66 | 11 | 19
titers | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.31 [4.69 to 6.01] | 5.17 [4.83 to 5.53] | 11.5 [6.17 to 21.4] | 17.4 [12.1 to 25.0] | 31.2 [16.4 to 59.4] | 69.0 [48.3 to 98.5] | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 5.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

4. Primary Outcome: Geometric Mean Fold-rise (GMFR) of Serum Neutralization Antibody Titers at Day 22
Description: SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. Fold-rise was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (Day 22) and pre-vaccination (on Day 1) i.e., Day 22/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 22 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 17 | 67 | 22 | 68 | 13 | 22
ratio | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.05 [0.945 to 1.18] | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.06 [0.977 to 1.15] | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.12 [0.986 to 1.27] | 1.07 [0.924 to 1.24] | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

5. Primary Outcome: Geometric Mean Fold-rise of Serum Neutralization Antibody Titers at Day 36
Description: SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. Fold-rise was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (Day 36) and pre-vaccination (on Day 1) i.e., Day 36/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 36 (post-vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 16 | 59 | 20 | 65 | 11 | 19
ratio | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.06 [0.938 to 1.20] | 1.03 [0.966 to 1.11] | 2.42 [1.26 to 4.67] | 3.36 [2.33 to 4.85] | 6.24 [3.27 to 11.9] | 14.0 [9.78 to 20.1] | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1.00 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

6. Primary Outcome: Number of Participants With >=2-fold and >=4-fold Rise in Serum Neutralization Antibody Titers at Day 22
Description: SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. The fold rise (2-fold and 4-fold) was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (on Day 22) and pre-vaccination (on Day 1) i.e., Day 22/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 22 (post-vaccination)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 17 | 67 | 22 | 68 | 13 | 22
Participants
  >=2-fold rise | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 4 | 1 | 0
  >=4-fold rise | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0

7. Primary Outcome: Number of Participants With >=2-Fold and >=4-Fold Rise in Serum Neutralization Antibody Titer at Day 36
Description: SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. The fold rise (2-fold and 4-fold) was calculated as the ratio of titer values of neutralizing antibodies post-vaccination (on Day 36) and pre-vaccination (on Day 1) i.e., Day 36/Day 1.
Time Frame: Day 1 (pre-vaccination) and Day 36 (post-vaccination)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 16 | 59 | 20 | 65 | 11 | 19
Participants
  >=2-fold rise | 0 | 0 | 0 | 1 | 1 | 7 | 31 | 14 | 57 | 0 | 0
  >=4-fold rise | 0 | 0 | 0 | 1 | 0 | 5 | 22 | 14 | 49 | 0 | 0

8. Primary Outcome: Percentage of Participants Achieving Seroconversion Against SARS-CoV-2 Virus Antigens at Day 22
Description: Seroconversion was defined as participants with a Baseline (Day 1) titer value below lower limit of quantification (LLOQ) with a detectable neutralization antibody titer above assay LLOQ post vaccination (at Day 22). LLOQ of the neutralization assay was a titer of 10.
Time Frame: Day 22 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 17 | 67 | 22 | 68 | 13 | 22
percentage of participants | 0 [0 to 14.2] | 0 [0 to 16.8] | 0 [0 to 16.8] | 4.2 [0.1 to 21.1] | 0 [0 to 13.7] | 0 [0 to 19.5] | 3.0 [0.4 to 10.4] | 0 [0 to 15.4] | 5.9 [1.6 to 14.4] | 7.7 [0.2 to 36.0] | 0 [0 to 15.4]

9. Primary Outcome: Percentage of Participants Achieving Seroconversion Against SARS-CoV-2 Virus Antigens at Day 36
Description: Seroconversion was defined as participants with a Baseline (Day 1) titer value below LLOQ with a detectable neutralization antibody titer above assay LLOQ post vaccination (at Day 36). LLOQ of the neutralization assay was a titer of 10.
Time Frame: Day 36 (post-vaccination)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03: Participants received IM injection of SARS-CoV2 vaccine LD formulation (5 mcg) along with adjuvant AS03 on Day 1 and Day 22, respectively.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 16 | 59 | 20 | 65 | 11 | 19
percentage of participants | 0 [0 to 15.4] | 0 [0 to 16.1] | 0 [0 to 17.6] | 4.2 [0.1 to 21.1] | 4.2 [0.1 to 21.1] | 43.8 [19.8 to 70.1] | 52.5 [39.1 to 65.7] | 70.0 [45.7 to 88.1] | 87.7 [77.2 to 94.5] | 0 [0 to 28.5] | 0 [0 to 17.6]

10. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessary had to have a causal relationship with treatment. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions prelisted in the case report form (CRF) in terms of diagnosis and/or onset window post-vaccination. All participants were observed for 30 minutes after vaccination, and any unsolicited systemic AEs occurred during that time were recorded as immediate unsolicited AEs in the CRF. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 30 minutes post any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 22])
Population: Analyzed on safety analysis set (SafAS) population which included randomized participants who had received at least one injection of study intervention and were analyzed according to study intervention they actually received. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were evaluable for assessment for the specified Group, as there was only 1 vaccination administered to Cohort 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 35 | 34 | 34 | 26 | 80 | 26 | 85 | 18 | 29
Participants
  Post any vaccination | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post vaccination 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 80 | 26 | 85 | 17 | 29
  Post vaccination 2 |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction (SR) was defined as an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRF and considered as related to vaccination. Solicited injection site reactions included pain, erythema and swelling. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days post any and each vaccination (Vaccination 1 [i.e., at Day 1] and 2 [i.e., at Day 22])
Population: Analysis was performed on SafAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM and 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were available for assessment for the specified Group, as there was only 1 vaccination administered to Cohort 1.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Group 10: SARS-CoV-2 Vaccine HD: Participants received IM injection of SARS-CoV2 vaccine LD formulation without adjuvant on Day 1 and Day 22, respectively.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 34 | 34 | 33 | 26 | 79 | 26 | 85 | 18 | 29
Participants
  Pain post-any vaccination | 18 | 30 | 21 | 28 | 5 | 19 | 73 | 20 | 80 | 4 | 6
  Pain post-vaccination 1 | 18 | 30 | 21 | 28 | 5 | 16 | 53 | 13 | 64 | 2 | 4
  Pain post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 79 | 26 | 85 | 17 | 29
  Pain post-vaccination 2 |  |  |  |  |  | 19 | 70 | 19 | 78 | 2 | 3
  Erythema post-any vaccination | 2 | 0 | 0 | 3 | 0 | 3 | 19 | 4 | 39 | 1 | 1
  Erythema post-vaccination 1 | 2 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 4 | 0 | 0
  Erythema post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 79 | 26 | 85 | 17 | 28
  Erythema post-vaccination 2 |  |  |  |  |  | 2 | 19 | 4 | 37 | 1 | 1
  Swelling post-any vaccination | 1 | 2 | 1 | 2 | 0 | 3 | 16 | 4 | 27 | 1 | 0
  Swelling post-vaccination 1 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 5 | 0 | 0
  Swelling post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 79 | 26 | 85 | 17 | 29
  Swelling post-vaccination 2 |  |  |  |  |  | 3 | 15 | 4 | 26 | 1 | 0

12. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: An SR was defined as an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the protocol and CRF and considered as related to vaccination. Solicited systemic reactions included fever, headache, malaise and myalgia. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 7 days post any and each vaccination (Vaccination 1 [i.e., Day 1] and 2 [i.e., Day 22])
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 34 | 34 | 33 | 26 | 80 | 26 | 85 | 18 | 29
Participants
  Fever post-any vaccination: number analyzed (Participants) | 35 | 36 | 34 | 34 | 32 | 26 | 80 | 26 | 85 | 18 | 29
  Fever post-any vaccination | 0 | 0 | 0 | 0 | 0 | 4 | 28 | 5 | 25 | 0 | 0
  Fever post-vaccination 1: number analyzed (Participants) | 35 | 36 | 34 | 34 | 32 | 26 | 78 | 26 | 85 | 18 | 29
  Fever post-vaccination 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
  Fever post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 78 | 26 | 84 | 16 | 29
  Fever post-vaccination 2 |  |  |  |  |  | 4 | 28 | 5 | 23 | 0 | 0
  Headache post-any vaccination | 10 | 13 | 4 | 11 | 6 | 14 | 60 | 17 | 59 | 5 | 7
  Headache post-vaccination 1: number analyzed (Participants) | 36 | 36 | 34 | 34 | 33 | 26 | 79 | 26 | 85 | 18 | 29
  Headache post-vaccination 1 | 10 | 13 | 4 | 11 | 6 | 3 | 20 | 7 | 34 | 4 | 7
  Headache post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 80 | 26 | 85 | 17 | 29
  Headache post-vaccination 2 |  |  |  |  |  | 13 | 57 | 16 | 53 | 3 | 3
  Malaise post-any vaccination: number analyzed (Participants) | 36 | 36 | 34 | 34 | 33 | 26 | 79 | 26 | 85 | 18 | 29
  Malaise post-any vaccination | 6 | 11 | 9 | 8 | 5 | 15 | 61 | 19 | 68 | 1 | 6
  Malaise post-vaccination 1: number analyzed (Participants) | 36 | 36 | 34 | 34 | 33 | 26 | 79 | 26 | 85 | 18 | 29
  Malaise post-vaccination 1 | 6 | 11 | 9 | 8 | 5 | 4 | 16 | 6 | 24 | 1 | 5
  Malaise post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 79 | 26 | 85 | 17 | 29
  Malaise post-vaccination 2 |  |  |  |  |  | 13 | 59 | 18 | 64 | 0 | 3
  Myalgia post-any vaccination | 6 | 12 | 13 | 15 | 6 | 15 | 63 | 19 | 69 | 3 | 3
  Myalgia post-vaccination 1: number analyzed (Participants) | 36 | 36 | 34 | 34 | 33 | 26 | 79 | 26 | 85 | 18 | 29
  Myalgia post-vaccination 1 | 6 | 12 | 13 | 15 | 6 | 5 | 22 | 9 | 32 | 2 | 2
  Myalgia post-vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 80 | 26 | 85 | 17 | 29
  Myalgia post-vaccination 2 |  |  |  |  |  | 12 | 60 | 18 | 65 | 2 | 3

13. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessary had to have a causal relationship with treatment. An unsolicited AE was an observed AE that did not fulfill the conditions of solicited reactions prelisted in the CRF in terms of diagnosis and/or onset post-vaccination. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: Within 21 days post any and each vaccination (Vaccination 1 [i.e., Day 1] and 2 [i.e., Day 22])
Population: Analysis was performed on SafAS population. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were available for assessment for the specified Group, as there was only 1 vaccination administered to Cohort 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 35 | 34 | 34 | 26 | 80 | 26 | 85 | 18 | 29
Participants
  Post any vaccination | 10 | 9 | 9 | 10 | 8 | 13 | 34 | 11 | 50 | 5 | 9
  Post vaccination 1 | 10 | 9 | 9 | 10 | 8 | 3 | 13 | 8 | 26 | 3 | 7
  Post vaccination 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 26 | 80 | 26 | 85 | 17 | 29
  Post vaccination 2 |  |  |  |  |  | 11 | 29 | 5 | 39 | 4 | 3

14. Primary Outcome: Number of Participants With Medically Attended Adverse Events (MAAE)
Description: A MAAE were AEs with a new onset or a worsening of a condition that prompted the participant to seek unplanned medical advice at a physician's office (including phone contact or email) or emergency department. An AE was defined as any untoward medical occurrence in a participant who received study vaccine and does not necessarily had to have a causal relationship with treatment. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 1 up to 12 months post last vaccination (i.e., up to Day 366 for Cohort 1 and up to Day 387 for Cohort 2)
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 35 | 34 | 34 | 26 | 80 | 26 | 85 | 18 | 29
Participants | 5 | 3 | 4 | 5 | 4 | 8 | 11 | 6 | 7 | 1 | 2

15. Primary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 1 up to 12 months post last vaccination (i.e., up to Day 366 for Cohort 1 and up to Day 387 for Cohort 2)
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 35 | 34 | 34 | 26 | 80 | 26 | 85 | 18 | 29
Participants | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0

16. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate. Reported AEs for each arm were presented as pre-specified in the study protocol.
Time Frame: From Day 1 up to 12 months post last vaccination (i.e., up to Day 366 for Cohort 1 and up to Day 387 for Cohort 2)
Population: Analysis was performed on SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 36 | 36 | 35 | 34 | 34 | 26 | 80 | 26 | 85 | 18 | 29
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Laboratory Test Results Based on US FDA Toxicity Grading Guidance
Description: Laboratory tests included hemoglobin (male and female), above and below normal white blood cell, lymphocytes, neutrophils & eosinophils, platelet count, creatinine and blood urea nitrogen, hyponatremia & hypernatremia, hyperkalemia & hypokalemia, hyperglycemia (non-fasting), hypoproteinemia, alkaline phosphate, alanine aminotransferase, aspartate aminotransferase, bilirubin (with any increase in liver function test [LFT], bilirubin (normal in LFT), amylase & lipase, Urine: protein, glucose & blood. The US FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" was used for grading. As per the guidance, Grade 1 = mild, Grade 2 = moderate and Grade 3 = severe.
Time Frame: From Day 1 up to 8 days post last dose (i.e., up to Day 9 for Cohort 1 and up to Day 30 for Cohort 2)
Population: Analysis was performed on SafAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM and 'number analyzed' = participants with available data for each specified category. Reported data for each arm were presented as pre-specified in the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 26 | 85 | 18 | 28
Participants
  Hemoglobin: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Hemoglobin: Grade 1 | 0 | 0 | 0 | 1 | 2 | 1 | 5 | 1 | 5 | 1 | 4
  Hemoglobin: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Hemoglobin: Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hemoglobin: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Hemoglobin: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hemoglobin (Female): Grade 1: number analyzed (Participants) | 22 | 15 | 18 | 21 | 18 | 13 | 34 | 16 | 44 | 10 | 14
  Hemoglobin (Female): Grade 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 4 | 1 | 1
  Hemoglobin (Female): Grade 2: number analyzed (Participants) | 22 | 15 | 18 | 21 | 18 | 13 | 34 | 16 | 44 | 10 | 14
  Hemoglobin (Female): Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hemoglobin (Female): Grade 3: number analyzed (Participants) | 22 | 15 | 18 | 21 | 18 | 13 | 34 | 16 | 44 | 10 | 14
  Hemoglobin (Female): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hemoglobin (Male): Grade 1: number analyzed (Participants) | 12 | 17 | 16 | 12 | 15 | 13 | 44 | 9 | 41 | 8 | 14
  Hemoglobin (Male): Grade 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 3
  Hemoglobin (Male): Grade 2: number analyzed (Participants) | 12 | 17 | 16 | 12 | 15 | 13 | 44 | 9 | 41 | 8 | 14
  Hemoglobin (Male): Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin (Male): Grade 3: number analyzed (Participants) | 12 | 17 | 16 | 12 | 15 | 13 | 44 | 9 | 41 | 8 | 14
  Hemoglobin (Male): Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Above normal white blood cell: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Above normal white blood cell: Grade 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Above normal white blood cell: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Above normal white blood cell: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Above normal white blood cell: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Above normal white blood cell: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Below normal white blood cell: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Below normal white blood cell: Grade 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Below normal white blood cell: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Below normal white blood cell: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Below normal white blood cell: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Below normal white blood cell: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Lymphocytes Decreased: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Lymphocytes Decreased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Lymphocytes Decreased: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Lymphocytes Decreased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Lymphocytes Decreased: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Lymphocytes Decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Neutrophils Decreased: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Neutrophils Decreased: Grade 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 5 | 0 | 2
  Absolute Neutrophils Decreased: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Neutrophils Decreased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Neutrophils Decreased: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Neutrophils Decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Eosinophils: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Eosinophils: Grade 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Absolute Eosinophils: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Eosinophils: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Absolute Eosinophils: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 84 | 17 | 28
  Absolute Eosinophils: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decreased: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Platelets Decreased: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets Decreased: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Platelets Decreased: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets Decreased: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 78 | 25 | 85 | 18 | 28
  Platelets Decreased: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Creatinine: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Grade 1 | 2 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 3 | 0 | 0
  Blood Urea Nitrogen: Grade 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1
  Blood Urea Nitrogen: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Hyponatremia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
  Hyponatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 77 | 26 | 85 | 18 | 28
  Hyperkalemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 77 | 26 | 85 | 18 | 28
  Hyperkalemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 77 | 26 | 85 | 18 | 28
  Hyperkalemia: Grade 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 77 | 26 | 85 | 18 | 28
  Hypokalemia: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 77 | 26 | 85 | 18 | 28
  Hypokalemia: Grade 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 3: number analyzed (Participants) | 34 | 32 | 34 | 33 | 33 | 26 | 77 | 26 | 85 | 18 | 28
  Hypokalemia: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia: Grade 1: number analyzed (Participants) | 31 | 32 | 33 | 31 | 33 | 23 | 71 | 25 | 78 | 18 | 27
  Hyperglycemia: Grade 1 | 2 | 3 | 1 | 1 | 6 | 0 | 2 | 0 | 4 | 1 | 2
  Hyperglycemia: Grade 2: number analyzed (Participants) | 31 | 32 | 33 | 31 | 33 | 23 | 71 | 25 | 78 | 18 | 27
  Hyperglycemia: Grade 2 | 2 | 0 | 1 | 0 | 0 | 0 | 5 | 0 | 3 | 1 | 2
  Hyperglycemia: Grade 3: number analyzed (Participants) | 31 | 32 | 33 | 31 | 33 | 23 | 71 | 25 | 78 | 18 | 27
  Hyperglycemia: Grade 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoproteinemia: Grade 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Hypoproteinemia: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoproteinemia: Grade 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphate: Grade 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Alkaline phosphate: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline phosphate: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase: Grade 1 | 2 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 3 | 2 | 2
  Alanine aminotransferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase: Grade 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 2 | 1 | 1
  Aspartate aminotransferase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin - with any increase in LFT: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin - with any increase in LFT: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Bilirubin - with any increase in LFT: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin - with normal in LFT: Grade 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Bilirubin - with normal in LFT: Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Bilirubin - with normal in LFT: Grade 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase: Grade 1 | 0 | 0 | 1 | 3 | 0 | 3 | 3 | 1 | 1 | 1 | 1
  Amylase: Grade 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Amylase: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase: Grade 1 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 2 | 0 | 1
  Lipase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lipase: Grade 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Urine - protein: Grade 1: number analyzed (Participants) | 33 | 32 | 34 | 33 | 32 | 26 | 78 | 26 | 85 | 18 | 28
  Urine - protein: Grade 1 | 2 | 3 | 4 | 1 | 2 | 1 | 9 | 4 | 10 | 2 | 2
  Urine - protein: Grade 2: number analyzed (Participants) | 33 | 32 | 34 | 33 | 32 | 26 | 78 | 26 | 85 | 18 | 28
  Urine - protein: Grade 2 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine - protein: Grade 3: number analyzed (Participants) | 33 | 32 | 34 | 33 | 32 | 26 | 78 | 26 | 85 | 18 | 28
  Urine - protein: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urine - glucose: Grade 1: number analyzed (Participants) | 33 | 32 | 34 | 33 | 32 | 26 | 78 | 26 | 85 | 18 | 28
  Urine - glucose: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine - glucose: Grade 2: number analyzed (Participants) | 33 | 32 | 34 | 33 | 32 | 26 | 78 | 26 | 85 | 18 | 28
  Urine - glucose: Grade 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine - glucose: Grade 3: number analyzed (Participants) | 33 | 32 | 34 | 33 | 32 | 26 | 78 | 26 | 85 | 18 | 28
  Urine - glucose: Grade 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Urine - blood: Grade 1: number analyzed (Participants) | 6 | 8 | 6 | 3 | 8 | 2 | 17 | 2 | 19 | 2 | 3
  Urine - blood: Grade 1 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Urine - blood: Grade 2: number analyzed (Participants) | 6 | 8 | 6 | 3 | 8 | 2 | 17 | 2 | 19 | 2 | 3
  Urine - blood: Grade 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
  Urine - blood: Grade 3: number analyzed (Participants) | 6 | 8 | 6 | 3 | 8 | 2 | 17 | 2 | 19 | 2 | 3
  Urine - blood: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Geometric Mean Concentration (GMC) of Anti-S Binding Antibody at Day 1, 22, 36, 181, 202, 366 and 387
Description: GMC of Anti-S binding antibodies were assessed using enzyme-linked immunosorbent assay (ELISA) and were measured in binding antibody units/milliliter (BAU/mL).
Time Frame: Day 1 (pre-vaccination); Day 22 (post-vaccination), Day 36 (post-vaccination), Day 181 (only for Cohort 1), Day 202 (only for Cohort 2), Day 366 (only for Cohort 1), and Day 387 (only for Cohort 2)
Population: Analysis was performed on PPAS-IAS population. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were evaluable for assessment in the specified Group for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/mL
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 21 | 20 | 24 | 25 | 18 | 68 | 22 | 69 | 13 | 22
BAU/mL
  Day 1: number analyzed (Participants) | 24 | 21 | 20 | 24 | 25 | 17 | 67 | 22 | 68 | 13 | 22
  Day 1 | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 9.80 [9.08 to 10.6] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 10.1 [8.76 to 11.8] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 11.7 [8.56 to 15.9] | 9.66 [9.25 to 10.1] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 9.73 [9.18 to 10.3] | 10.5 [8.34 to 13.3] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Day 22: number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 17 | 68 | 22 | 69 | 13 | 22
  Day 22 | 34.7 [18.8 to 63.8] | 61.8 [35.8 to 107] | 46.1 [24.8 to 86.0] | 160 [78.4 to 327] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 45.2 [21.0 to 97.0] | 88.4 [60.6 to 129] | 50.2 [28.6 to 88.4] | 136 [101 to 184] | 10.4 [8.44 to 12.8] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Day 36: number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 17 | 60 | 20 | 66 | 11 | 19
  Day 36 | 26.0 [13.9 to 48.8] | 73.7 [43.2 to 126] | 41.0 [22.2 to 75.5] | 136 [70.2 to 264] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 1049 [448 to 2457] | 3571 [2597 to 4910] | 3086 [1781 to 5346] | 7842 [6120 to 10049] | 29.8 [15.4 to 57.4] | 9.45 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Day 181: number analyzed (Participants) | 15 | 14 | 11 | 14 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181 | 50.9 [15.0 to 172] | 145 [27.8 to 757] | 21.7 [11.2 to 42.2] | 127 [21.1 to 765] | 44.6 [9.75 to 204] |  |  |  |  |  |
  Day 202: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 26 | 8 | 27 | 4 | 5
  Day 202 |  |  |  |  |  | 925 [2.78 to 307000] | 828 [344 to 1993] | 1338 [154 to 11655] | 3451 [1439 to 8275] | 28070 [7802 to 101000] | 217 [4.01 to 11732]
  Day 366: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366 | 2161 [92.8 to 50304] | 7355 [221 to 245000] | 1250 [126 to 12379] | 12580 [2121 to 74606] | 6265 [361 to 109000] |  |  |  |  |  |
  Day 387: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 10 | 6 | 10 | 2 | 1
  Day 387 |  |  |  |  |  | 3439 [0 to 1000000] | 9009 [738 to 110000] | 24115 [10016 to 58060] | 37532 [13416 to 105000] | 4114 [0.641 to 26400000] | 1126 [NA to NA] — 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

19. Secondary Outcome: Geometric Mean Fold-rise (GMFR) of Binding Antibody Concentration at Day 22, 36, 181, 202, 366 and 387
Description: Binding antibody titers were evaluated by ELISA. Fold-rise was calculated as the ratio of geometric mean concentrations of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., Day 22/Day 01, Day 36/Day 01, Day 181/Day 1, Day 202/Day 1, Day 366/Day 1, and Day 387/Day 1.
Time Frame: as for outcome 18
Population: Analysis was performed on PPAS-IAS population. Here, "overall number of participants analyzed" signifies participants with available data for this OM, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field denotes that none of the participants were evaluable for assessment in the specified Group for the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 21 | 20 | 24 | 25 | 17 | 67 | 22 | 68 | 13 | 22
ratio
  Day 22/Day 1: number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 16 | 67 | 22 | 68 | 13 | 22
  Day 22/Day 1 | 3.67 [1.99 to 6.76] | 6.30 [3.69 to 10.8] | 4.88 [2.62 to 9.10] | 15.8 [8.08 to 30.8] | 1.00 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 3.67 [1.85 to 7.28] | 9.12 [6.24 to 13.3] | 5.32 [3.02 to 9.36] | 13.8 [10.2 to 18.7] | 0.989 [0.966 to 1.01] | 1.00 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Day 36/Day 1: number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 16 | 59 | 20 | 65 | 11 | 19
  Day 36/Day 1 | 2.75 [1.47 to 5.16] | 7.52 [4.45 to 12.7] | 4.34 [2.35 to 7.99] | 13.4 [7.18 to 25.1] | 1.00 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 91.0 [36.6 to 226] | 367 [267 to 504] | 327 [188 to 566] | 812 [621 to 1061] | 2.78 [1.34 to 5.75] | 1.00 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.
  Day 181/Day 1: number analyzed (Participants) | 15 | 14 | 11 | 14 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1 | 5.39 [1.59 to 18.2] | 14.5 [2.76 to 76.3] | 2.30 [1.18 to 4.47] | 13.4 [2.23 to 80.9] | 4.72 [1.03 to 21.6] |  |  |  |  |  |
  Day 202/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202/Day 1 |  |  |  |  |  | 58.2 [0.910 to 3722] | 68.9 [30.3 to 156] | 142 [16.2 to 1233] | 387 [157 to 954] | 2970 [826 to 10687] | 23.0 [0.424 to 1241]
  Day 366/Day 1: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366/Day 1 | 229 [9.82 to 5323] | 685 [21.0 to 22298] | 132 [13.4 to 1310] | 1331 [224 to 7895] | 663 [38.2 to 11509] |  |  |  |  |  |
  Day 387/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1 |  |  |  |  |  | 364 [0 to 1000000] | 933 [53.9 to 16147] | 2552 [1060 to 6144] | 3972 [1420 to 11111] | 435 [0.068 to 2800000] | 119 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

20. Secondary Outcome: Number of Participants With >=2-Fold and >=4- Fold Rise in Anti-S Binding Antibody Concentration at Day 22, 36, 181, 202, 366 and 387
Description: Binding Antibody Titers were evaluated by ELISA. Fold rise (2-fold and 4-fold) was calculated as the ratio of titer values for binding antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., Day 22/Day 1 and Day 36/Day 1, Day 181/Day 1, Day 202/Day 1, Day 366/Day 1, and Day 387/Day 1.
Time Frame: as for outcome 18
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 24 | 21 | 20 | 24 | 25 | 18 | 67 | 22 | 68 | 13 | 22
Participants
  Day 22/Day 1: >=2-fold rise: number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 16 | 67 | 22 | 68 | 13 | 22
  Day 22/Day 1: >=2-fold rise | 14 | 17 | 15 | 21 | 0 | 10 | 55 | 17 | 66 | 0 | 0
  Day 22/Day 1: >=4-fold rise: number analyzed (Participants) | 24 | 20 | 20 | 24 | 25 | 16 | 67 | 22 | 68 | 13 | 22
  Day 22/Day 1: >=4-fold rise | 10 | 12 | 9 | 18 | 0 | 8 | 46 | 13 | 56 | 0 | 0
  Day 36/Day 1: >=2-fold rise: number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 16 | 59 | 20 | 65 | 11 | 19
  Day 36/Day 1: >=2-fold rise | 9 | 18 | 14 | 21 | 0 | 15 | 59 | 20 | 65 | 7 | 0
  Day 36/Day 1: >=4-fold rise: number analyzed (Participants) | 22 | 21 | 19 | 24 | 24 | 16 | 59 | 20 | 65 | 11 | 19
  Day 36/Day 1: >=4-fold rise | 8 | 15 | 9 | 20 | 0 | 15 | 58 | 20 | 65 | 3 | 0
  Day 181/Day 1: >=2-fold rise: number analyzed (Participants) | 15 | 14 | 11 | 14 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=2-fold rise | 10 | 11 | 6 | 11 | 4 |  |  |  |  |  |
  Day 181/Day 1: >=4-fold rise: number analyzed (Participants) | 15 | 14 | 11 | 14 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=4-fold rise | 6 | 10 | 3 | 7 | 4 |  |  |  |  |  |
  Day 202/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202/Day 1: >=2-fold rise |  |  |  |  |  | 4 | 25 | 8 | 26 | 4 | 3
  Day 202/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202/Day 1: >=4-fold rise |  |  |  |  |  | 4 | 25 | 8 | 26 | 4 | 3
  Day 366/Day 1: >=2-fold rise: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366/Day 1: >=2-fold rise | 5 | 5 | 6 | 7 | 6 |  |  |  |  |  |
  Day 366/Day 1: >=4-fold rise: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366/Day 1: >=4-fold rise | 5 | 5 | 6 | 7 | 6 |  |  |  |  |  |
  Day 387/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1: >=2-fold rise |  |  |  |  |  | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1: >=4-fold rise |  |  |  |  |  | 2 | 8 | 6 | 10 | 2 | 1

21. Secondary Outcome: Geometric Mean Titers of Neutralizing Antibodies Against SARS-CoV-2 Recombinant Protein Vaccine Formulations at Day 181, 202, 366 and 387
Description: as for outcome 1
Time Frame: Cohort 1: Day 181 and Day 366 and Cohort 2: Day 202 and Day 387 (post-vaccination)
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 4 | 26 | 8 | 27 | 4 | 5
titers
  Day 181: number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181 | 6.89 [3.91 to 12.2] | 8.81 [3.74 to 20.7] | 5.00 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 9.99 [3.62 to 27.5] | 10.9 [4.73 to 25.3] |  |  |  |  |  |
  Day 202: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 26 | 8 | 27 | 4 | 5
  Day 202 |  |  |  |  |  | 31.7 [0.089 to 11282] | 14.5 [6.47 to 32.4] | 30.8 [3.50 to 271] | 53.6 [21.3 to 135] | 355 [84.7 to 1486] | 16.0 [2.18 to 117]
  Day 366: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366 | 35.6 [6.67 to 190] | 159 [21.2 to 1199] | 36.3 [3.51 to 376] | 127 [29.3 to 551] | 242 [33.4 to 1761] |  |  |  |  |  |
  Day 387: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 10 | 6 | 10 | 2 | 1
  Day 387 |  |  |  |  |  | 30.1 [0 to 240000000000] | 235 [28.8 to 1913] | 727 [361 to 1465] | 1043 [324 to 3355] | 39.7 [0.006 to 245000] | 23.0 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

22. Secondary Outcome: Geometric Mean Fold-rise of Serum Neutralization Antibody Titer at Day 181, 202, 366 and 387
Description: SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. Fold-rise was calculated as the ratio of titer values of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., for Cohort 1: Day 181/Day 1 and Day 366/Day 1; Cohort 2: Day 202/Day 1 and Day 387/Day 1.
Time Frame: Day 1 (pre-vaccination), Cohort 1: Day 181 and Day 366 and Cohort 2: Day 202 and Day 387 (post-vaccination)
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 4 | 25 | 8 | 26 | 4 | 5
ratio
  Day 181/Day 1: number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1 | 1.38 [0.781 to 2.43] | 1.76 [0.748 to 4.15] | 1.00 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value. | 2.00 [0.724 to 5.51] | 2.19 [0.947 to 5.05] |  |  |  |  |  |
  Day 202/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202/Day 1 |  |  |  |  |  | 6.34 [0.018 to 2256] | 2.38 [1.15 to 4.91] | 6.16 [0.699 to 54.3] | 11.7 [4.59 to 30.1] | 71.0 [16.9 to 297] | 3.20 [0.436 to 23.5]
  Day 366/Day 1: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366/Day 1 | 7.12 [1.33 to 38.0] | 31.9 [4.23 to 240] | 7.26 [0.701 to 75.2] | 25.4 [5.86 to 110] | 48.5 [6.67 to 352] |  |  |  |  |  |
  Day 387/Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1 |  |  |  |  |  | 6.02 [0 to 1000000] | 49.5 [4.55 to 539] | 145 [72.2 to 293] | 209 [64.8 to 671] | 7.95 [0.001 to 49046] | 4.60 [NA to NA] — NA Explanation: 95% CI was not computable as the SD of the sample was 0, since all participants had the same value.

23. Secondary Outcome: Number of Participants With 2-Fold and 4-Fold Rise in Serum Neutralization Antibody Titer at Day 181, 202, 366 and 387
Description: SARS-CoV-2 neutralizing antibodies was measured using a neutralization assay. The fold rise (2-fold and 4-fold) was calculated as the ratio of titer values of antibodies post-vaccination at specified timepoints and pre-vaccination (on Day 1) i.e., Cohort 1: Day 181/Day 1 and Day 366/Day 1 and Cohort 2: Day 202/Day 1 and Day 387/Day 1.
Time Frame: Day 1 (pre-vaccination), Cohort 1: Day 181 and Day 366 and Cohort 2: Day 202 and Day 387 (post-vaccination)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 4 | 25 | 8 | 26 | 4 | 5
Participants
  Day 181/Day 1: >=2-fold rise: number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=2-fold rise | 2 | 2 | 0 | 2 | 4 |  |  |  |  |  |
  Day 202/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202/Day 1: >=2-fold rise |  |  |  |  |  | 1 | 6 | 3 | 19 | 4 | 2
  Day 181/Day 1: >=4-fold rise: number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181/Day 1: >=4-fold rise | 1 | 2 | 0 | 2 | 3 |  |  |  |  |  |
  Day 202/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202/Day 1: >=4-fold rise |  |  |  |  |  | 1 | 5 | 3 | 14 | 4 | 2
  Day 366/Day 1: >=2-fold rise: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366/Day 1: >=2-fold rise | 4 | 5 | 3 | 6 | 6 |  |  |  |  |  |
  Day 387/Day 1: >=2-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1: >=2-fold rise |  |  |  |  |  | 1 | 7 | 6 | 10 | 2 | 1
  Day 366/Day 1: >=4-fold rise: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366/Day 1: >=4-fold rise | 3 | 5 | 3 | 6 | 6 |  |  |  |  |  |
  Day 387/Day 1: >=4-fold rise: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387/Day 1: >=4-fold rise |  |  |  |  |  | 1 | 6 | 6 | 10 | 2 | 1

24. Secondary Outcome: Percentage of Participants Achieving Seroconversion Against SARS-CoV2 Virus Antigens at Day 181, 202, 366 and 387
Description: Seroconversion was defined as participants with a Baseline (Day 1) titer value below LLOQ with a detectable neutralization antibody titer above assay LLOQ post vaccination (Cohort 1: Day 181 and Day 366 and Cohort 2: Day 202 and Day 387). LLOQ of the neutralization assay was a titer of 10.
Time Frame: Cohort 1: Day 181 and Day 366 and Cohort 2: Day 202 and Day 387 (post-vaccination)
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 4 | 25 | 8 | 26 | 4 | 5
percentage of participants
  Day 181: number analyzed (Participants) | 15 | 14 | 11 | 15 | 16 | 0 | 0 | 0 | 0 | 0 | 0
  Day 181 | 13.3 [1.7 to 40.5] | 14.3 [1.8 to 42.8] | 0 [0 to 28.5] | 13.3 [1.7 to 40.5] | 25.0 [7.3 to 52.4] |  |  |  |  |  |
  Day 202: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 25 | 8 | 26 | 4 | 5
  Day 202 |  |  |  |  |  | 25.0 [0.6 to 80.6] | 24.0 [9.4 to 45.1] | 37.5 [8.5 to 75.5] | 73.1 [52.2 to 88.4] | 100 [39.8 to 100] | 40.0 [5.3 to 85.3]
  Day 366: number analyzed (Participants) | 5 | 6 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0
  Day 366 | 80.0 [28.4 to 99.5] | 83.3 [35.9 to 99.6] | 50.0 [11.8 to 88.2] | 85.7 [42.1 to 99.6] | 85.7 [42.1 to 99.6] |  |  |  |  |  |
  Day 387: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2 | 9 | 6 | 10 | 2 | 1
  Day 387 |  |  |  |  |  | 50.0 [1.3 to 98.7] | 77.8 [40.0 to 97.2] | 100 [54.1 to 100] | 100 [69.2 to 100] | 100 [15.8 to 100] | 100 [2.5 to 100]

25. Secondary Outcome: Number of Participants With Virologically-confirmed Coronavirus Disease (COVID-19)-Like Illness
Description: Virologically-confirmed COVID-19-like illness was defined by specified clinical symptoms and signs and confirmed by positive result for SARS-CoV-2 by nucleic acid amplification test (NAAT) on a respiratory sample in association with a COVID-19-like illness. The various COVID-19-like illness symptoms were cough, fever, anosmia, ageusia, chillblains, difficulty breathing, shortness of breath, pneumonia, stroke, myocarditis, myocardial infarction, thromboembolic event, purpura fulminans, pharyngitis, chills, myalgia, headache, rhinorrhea, abdominal pain, nausea, diarrhea and vomiting.
Time Frame: Cohort 1: up to Day 366 (post-vaccination) and Cohort 2: up to Day 387 (post-vaccination)
Population: Data for this OM (virologically confirmed COVID-19 like illness) was not collected and analyzed because of the limited number of COVID-19 cases before receiving an authorized/approved COVID-19 vaccine, and thus the corresponding anti-nucleoprotein testing was not conducted, and the planned efficacy analysis was not performed.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Serologically-confirmed SARS-CoV-2 Infection
Description: Serologically-confirmed SARS-CoV-2 infection was defined as a change from negative to positive result in serum for presence of antibodies specific to non-Spike protein of SARS-CoV-2 detected by ELISA assay from any post-baseline sampling time point compared to the Baseline value.
Time Frame: Cohort 1: up to Day 366 (post-vaccination) and Cohort 2: up to Day 387 (post-vaccination)
Population: Data for this OM (serologically confirmed SARS-CoV2 infection) was not collected and analyzed because of the limited number of COVID-19 cases before receiving an authorized/approved COVID-19 vaccine, and thus the corresponding anti-nucleoprotein testing was not conducted, and the planned efficacy analysis was not performed.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Correlates of Risk / Protection Based on Antibody Responses to SARS-CoV-2
Description: Correlate of risk / protection based on antibody responses to SARS-CoV-2 was evaluated using virus neutralization or ELISA, considering virologically-confirmed COVID-19-like illness and/or serologically-confirmed SARS-CoV-2 infection.
Time Frame: From Day 1 up to Day 366 for Cohort 1 and up to Day 387 for Cohort 2
Population: Data for this OM (Correlates of Risk / Protection Based on Antibody Responses to SARS-CoV-2) was not collected and analyzed because of the limited number of COVID-19 cases before receiving an authorized/approved COVID-19 vaccine, and thus the corresponding anti-nucleoprotein testing was not conducted, and the planned efficacy analysis was not performed.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AE: from Day 0 (pre-vaccination) up to 21 days post any vaccination. Solicited reactions: collected within 7 days post any vaccination. SAE data were collected from Day 1 up to 12 months post last vaccination (i.e., up to Day 366 for Cohort 1 and up to Day 387 for Cohort 2)
Description: SR: defined as an "expected" AR (sign or symptom) observed and reported under conditions prelisted (i.e., solicited) in protocol and CRF and considered as related to vaccination. Unsolicited AE: an observed AE that did not fulfill conditions of solicited reactions prelisted in the CRF in terms of diagnosis and/or onset window post-vaccination. SafAS population. In AE section, solicited reaction Fever was reported as Pyrexia. Reported AEs for each arm were presented as pre-specified in protocol.
Arm/Group | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 | Cohort 1: Group 5: Placebo | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD | Cohort 2: Group 11: Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/35 | 0/34 | 0/34 | 0/26 | 0/80 | 0/26 | 0/85 | 0/18 | 0/29
Serious Adverse Events (participants affected / at risk) | 2/36 | 1/36 | 1/35 | 0/34 | 0/34 | 1/26 | 1/80 | 0/26 | 2/85 | 0/18 | 0/29
Other Adverse Events (participants affected / at risk) | 22/36 | 31/36 | 23/35 | 31/34 | 15/34 | 21/26 | 75/80 | 25/26 | 84/85 | 10/18 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 (N=36) | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 (N=36) | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 (N=35) | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 (N=34) | Cohort 1: Group 5: Placebo (N=34) | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 (N=26) | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 (N=80) | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 (N=26) | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 (N=85) | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD (N=18) | Cohort 2: Group 11: Placebo (N=29)
Nipple Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Group 1: SARS-CoV-2 Vaccine LD + AF03 (N=36) | Cohort 1: Group 2: SARS-CoV-2 Vaccine LD + AS03 (N=36) | Cohort 1: Group 3: SARS-CoV-2 Vaccine HD + AF03 (N=35) | Cohort 1: Group 4: SARS-CoV-2 Vaccine HD + AS03 (N=34) | Cohort 1: Group 5: Placebo (N=34) | Cohort 2: Group 6: SARS-CoV-2 Vaccine LD + AF03 (N=26) | Cohort 2: Group 7: SARS-CoV-2 Vaccine LD + AS03 (N=80) | Cohort 2: Group 8: SARS-CoV-2 Vaccine HD + AF03 (N=26) | Cohort 2: Group 9: SARS-CoV-2 Vaccine HD + AS03 (N=85) | Cohort 2: Group 10: SARS-CoV-2 Vaccine HD (N=18) | Cohort 2: Group 11: Placebo (N=29)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (9) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (7) | 2 (2) | 7 (8) | 1 (1) | 2 (2)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 13 (14) | 1 (1) | 10 (11) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Injection Site Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection Site Erythema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 19 (20) | 4 (5) | 39 (41) | 1 (1) | 1 (1)
Injection Site Pain (General disorders) | 18 (18) | 30 (30) | 21 (21) | 28 (28) | 5 (5) | 19 (35) | 73 (123) | 20 (32) | 80 (142) | 4 (4) | 6 (7)
Injection Site Pruritus (General disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 16 (18) | 0 (0) | 0 (0)
Injection Site Swelling (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 16 (16) | 4 (4) | 27 (31) | 1 (1) | 0 (0)
Malaise (General disorders) | 6 (6) | 12 (12) | 9 (9) | 8 (8) | 5 (5) | 15 (17) | 61 (75) | 19 (24) | 68 (88) | 1 (1) | 6 (8) — Malaise event which occurred 7 days post-vaccination was considered as an unsolicited AE.
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 28 (30) | 7 (8) | 25 (25) | 0 (0) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 12 (12) | 13 (13) | 16 (16) | 6 (6) | 16 (18) | 63 (85) | 19 (28) | 69 (98) | 3 (4) | 3 (5) — Myalgia events which occurred 7 days post-vaccination was considered as an unsolicited AE.
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 10 (10) | 13 (13) | 4 (4) | 11 (12) | 7 (7) | 14 (18) | 60 (81) | 18 (26) | 61 (91) | 6 (10) | 7 (11) — Headache events which occurred 7 days post-vaccination was considered as an unsolicited AE.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the limited number of COVID-19 cases before receiving an authorized/approved COVID-19 vaccine, the corresponding anti-nucleoprotein testing was not conducted, the planned few efficacy outcome measures data were not collected and analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT04537208/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04537208/SAP_001.pdf